CLINICAL TRIAL: NCT00956956
Title: A Phase I, Randomized, Placebo Controlled, Multiple Dose Study To Determine Safety, Tolerability And Pharmacokinetics Of PF-04455242 In Healthy Adult Subjects
Brief Title: A Multiple Dose Study To Determine Safety, Tolerability And Pharmacokinetics Of PF-04455242 In Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: B1071002
Record Dates: First submitted 2009-08-10; First posted 2009-08-11 (Estimated); Last update posted 2010-01-07 (Estimated); Status verified 2010-01

CONDITIONS: Healthy
Keywords: An investigator and subject blinded (sponsor open); multiple dose; dose escalation design with PF 04455242 and matching placebo.
MeSH Terms: interventions — 2-methyl-N-((2'-(pyrrolidin-1-ylsulfonyl)biphenyl-4-yl)methyl)propan-1-amine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PF-04455242 treatment (Experimental)
  Interventions: Drug: PF-04455242
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-04455242 — 3, 6, and 23 mg capsules administered orally Q6 hours for 7 days of dosing.
  Arms: PF-04455242 treatment
Drug: Placebo — Placebo administered orally Q6 hours for 7 days of dosing.
  Arms: Placebo

SUMMARY:
The goals of this study are to evaluate the safety and tolerability of multiple ascending doses of PF-04455242 administered orally to healthy adult subjects. In addition, the plasma and urine pharmacokinetics of multiple ascending doses of PF 04455242 administered orally to healthy adult subjects will be evaluated. Finally, the effect of multiple-doses of PF-04455242 on serum prolactin concentration will be explored.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects without childbearing potential between the ages of 21 and 55 years, inclusive. (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12 lead ECG and clinical laboratory tests).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies).

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2009-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of multiple ascending doses of PF 04455242 administered orally to healthy adult subjects. | 10 days
Plasma and urine pharmacokinetics of multiple ascending doses of PF 04455242 administered orally to healthy adult subjects. | 10 days

SECONDARY OUTCOMES:
Effect of multiple-doses of PF 04455242 on serum prolactin concentration. | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Singapore, Singapore

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1071002&StudyName=A%20Multiple%20Dose%20Study%20To%20Determine%20Safety%2C%20Tolerability%20And%20Pharmacokinetics%20Of%20PF-04455242%20In%20Healthy%20Adult%20Subjects